CLINICAL TRIAL: NCT00001734
Title: Screening Study for the Evaluation and Diagnosis of Potential Research Subjects With Ocular Inflammatory or Immunologic Diseases
Brief Title: Screening for NEI Clinical Studies
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980085; 98-EI-0085
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-03

CONDITIONS: Conjunctivitis; Iritis; Keratitis; Retinitis; Uveitis
Keywords: Uveitis; Conjunctivitis; Iritis; Retinitis; Keratitis; Screening Protocol; Ocular Immunology; Inflammation; Eye Inflammation
MeSH Terms: conditions — Conjunctivitis; Iritis; Keratitis; Retinitis; Uveitis; Inflammation; Endophthalmitis

SUMMARY:
This screening protocol is designed to facilitate patient recruitment to National Eye Institute (NEI) clinical research studies. Patients must meet specific requirements of a research study; this protocol serves as a first step for admitting patients to an appropriate program.

Candidates may have a diagnosed or undiagnosed eye condition. They will be screened with a medical history, physical examination, eye examination and blood test. Other screening procedures may include routine laboratory tests, non-invasive imaging, and questionnaires. The eye examination includes measurement of eye pressure and dilation of the pupils to fully examine the lens, vitreous and retina. Specialized eye tests will be done only if needed to determine eligibility for a specific study. When the screening is completed, patients will be informed of their options to participate in a study. Patients who are found ineligible for a current study will be informed of alternative treatments or options. No treatment is offered under this protocol.

DETAILED DESCRIPTION:
This protocol is designed for the screening of patients with either diagnosed or undiagnosed conditions, and serves as a first step for individuals who may be eligible, and wish to participate in NEI- National Eye Institute clinical research studies.

Each individual will be thoroughly evaluated during the screening process to determine if they are suitable candidates for inclusion in any of the NEI ongoing studies. The screening evaluation will include past and current medical histories, and an appropriate physical examination. Other routine diagnostic procedures and tests may also be completed in order to help determine a subject's eligibility. These tests and procedures are of minimal risk and will be described in more detail in section III: "Study Procedures". Once the screening process is completed and their eligibility is assessed, the subjects will be informed of their options to participate in one or more of the current clinical research studies. If no appropriate protocol is identified, recommendations for other treatment options may be given to the individual, their primary doctor, or referring physician.

ELIGIBILITY:
* Participants will be able to enroll if they:

  1. Have a diagnosed ocular inflammatory eye disease; OR
  2. Have an unusual, interesting or unknown ocular condition that requires the establishment of a diagnosis; AND
  3. Have the ability to understand and sign an informed consent OR have a legal parent/guardian with the ability to do the same.

2.2 Exclusion Criteria

Participants will be unable to enroll if they:

1. Have no ocular medical conditions; OR
2. Are unwilling or unable to cooperate with the procedures.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000
Dates: Start 1998-03-23; Study Completion 2008-10-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States